CLINICAL TRIAL: NCT00893659
Title: The Effect of Beta-glucan on Faecal Microflora in Polypectomized Patients
Brief Title: Beta-glucan on Fecal Microflora in Polypectomized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: JOTIS S.A. FOOD INDUSTRY, GREECE (Unknown)
Responsible Party: Principal Investigator, Kyriacou Adamantini, Assistant Professor, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HAR-GLUCAN-1
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Polypectomized Patients
Keywords: Beta-glucan; faecal microflora; polypectomized; Precancerous Nonmalignant Condition
MeSH Terms: interventions — beta-Glucans

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wheat bread with beta-glucan supplementation (Experimental)
  Interventions: Dietary Supplement: wheat bread with beta-glucan
- wheat bread without beta-glucan (Placebo Comparator)
  Interventions: Dietary Supplement: wheat bread without beta-glucan

INTERVENTIONS:
Dietary Supplement: wheat bread with beta-glucan — 3 g beta-glucan in approximately 200 g of wheat bread per day for 3 months
  Arms: wheat bread with beta-glucan supplementation
Dietary Supplement: wheat bread without beta-glucan — Approximately 200 g of wheat bread (without beta-glucan supplementation) per day for 3 months
  Arms: wheat bread without beta-glucan

SUMMARY:
The aim of this study is to determine the effect of the potential prebiotic beta-glucan on the intestinal microflora, the bacterial enzyme activity (beta-glucuronidase and beta-glucosidase) in the feces, the fecal pH and the concentration of fecal short-chain fatty acid in polypectomized patients. Also the in vitro anti-cyto- and anti-genotoxicity of fecal water will be examined on human cell culture (HT29). During the trial, patient's clinical symptoms (intestinal habits), physical activity, well-being and food intake will be recorded.

DETAILED DESCRIPTION:
Prebiotics, such as short- and long-chain fructo-oligosaccharides are fermented by the microflora colonizing the gastrointestinal tract, and they selectively stimulate the growth or the activity of one or limited number of bacteria within the intestine. Beta-glucans are polysaccharides occurring in the bran of cereal grains, the cell wall of Saccharomyces cerevisiae and bacteria, certain types of fungi, seaweed and many kinds of mushrooms. The aim of this study is to determine the effect of the potential prebiotic beta-glucan on the intestinal microflora, the bacterial enzyme activity (beta-glucuronidase and beta-glucosidase) in the faeces, the faecal pH, and the concentration of faecal short-chain fatty acid in polypectomized patients.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must have biopsy and histologically confirmed adenomatous polyps ≥ 1cm in size or ≥ 3 in number with moderate or severe dysplasia

Exclusion Criteria:

* Subjects ≥ 75 years of age
* Subjects who are pregnant or desire to become pregnant during the study period
* Subjects who are considered to be poor clinic attendees
* Subjects who have been on antibiotics within the previous month or are likely to require antibiotics during the trial
* Subjects who consume prebiotics or probiotics within the previous month or are likely to require antibiotics during the trial
* Subjects with colon cancer
* Subjects with additional gastrointestinal disorders (e.g., Crohn's disease or ulcerative colitis)
* Subjects with malignancy or any end-stage organ disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To measure the effect of beta-glucan on fecal microflora (number of bacteria, bacterial enzyme activity, SCFA, pH). | four months
To observe the effect of beta-glucan on intestinal symptoms and well-being. | four months

SECONDARY OUTCOMES:
To study the fecal water cyto- and/or genotoxicity on HT-29 cell line. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Adamantini Kyriacou, Ass. Professor, Study Director — Harokopio University
Locations (1):
- Harokopio University, Athens, Attica, Greece